CLINICAL TRIAL: NCT01650740
Title: A Randomized Trial of Sequenced Treatment Using Placebo Without Deception Followed by Open-Label Antidepressant Versus Immediate Open-Label Antidepressant Treatment for Major Depressive Disorder
Brief Title: Study of Placebo Without Deception Versus Standard Antidepressant for Major Depressive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment results.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 081-2012
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open-label duloxetine (Experimental): 12 week treatment with duloxetine
  Interventions: Drug: Duloxetine
- Open-label Placebo (Experimental): 4 weeks of open label placebo with option to continue or switch to duloxetine for remaining 8 weeks.
  Interventions: Drug: placebo
- Supportive clinical management (Experimental): 4 weeks of supportive clinical management visits with option to continue or switch to duloxetine for remaining 8 weeks.
  Interventions: Other: Study visits only

INTERVENTIONS:
Drug: Duloxetine — 30 mg daily x 1 week followed by 60 mg daily
  Other Names: cymbalta
  Arms: Open-label duloxetine
Drug: placebo — small placebo capsule (30 mg duloxetine equivalent) x 1 week followed by 60 mg equivalent capsule daily
  Arms: Open-label Placebo
Other: Study visits only — Weekly visits x 4 weeks followed by visits every 2 weeks
  Arms: Supportive clinical management

SUMMARY:
In recent years, there has been growing evidence that antidepressants are only marginally effective compared to placebo for mild to moderate depression. In other words, although many people improve when they take antidepressant medications, almost as many get better with placebo pills. One possible solution to this problem would be to give patients a trail of a placebo prior to giving them an antidepressant, however there are ethical issues with doing this deceptively. New evidence from other placebo-responsive disorders such as irritable bowel syndrome shows that people may benefit from placebos even if they know they are taking them. This study aims to determine whether giving placebos without deception to people with major depressive disorder followed by the option to switch to an antidepressant is an effective strategy. There will be 3 groups of subjects. The first group is a standard treatment arm and will receive duloxetine, an antidepressant. The second will be given a placebo with the option to switch to duloxetine if they do not improve. The third group will receive supportive clinical visits the option to switch to duloxetine if they do not improve. This design will allow us to determine whether a sequenced treatment of a placebo without deception and then the option to switch to an antidepressant is a viable strategy. It will also help us to determine to what degree the benefit comes from the ritual of receiving and taking the placebo tablet versus the benefit of visits with a doctor alone. The primary hypothesis is that there will be a less than 5% difference between response rates after 12 weeks in the sequenced placebo-then-antidepressant treatment group (both subjects who have remained on placebo as well as those who have switched to the antidepressant will be considered as one group) compared to the immediate antidepressant therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Diagnosis of major depressive disorder, currently depressed as determined by DSM-IV diagnostic criteria (confirmed using the MINI)
* Both females and males, aged 18 to 65 years
* Outpatient status
* Female patients of childbearing potential must have a negative urine human chorionic gonadotropin (hCG) test at enrolment and must be taking or willing to take some acceptable form of birth control during the course of the study if they are or plan to be sexually active
* A grade 8 English comprehension, the ability to understand and comply with the requirements of the study and capable of providing informed consent
* 17-item Hamilton Depression Rating Scale (HAM-D) score of 14-22 at screening and at baseline

Exclusion Criteria:

* Diagnosis of a past hypomanic, manic or mixed state.
* Current or past psychotic symptoms
* Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
* Any pervasive developmental disorder (according to DSM-IV criteria)
* Diagnosis of dementia (according to DSM-IV criteria)
* Is at significant risk for suicide, as defined by a score of ≥ 2 on the suicide item of the MADRS, any suicidal ideation with intent or a plan within the 3 months prior to study entry or in the opinion of the investigator.
* Any history of lifetime suicide attempts
* Current treatment with an antidepressant medication
* Treatment with an antipsychotic, mood stabilizer or other psychoactive medication within a period of 5 half-lives of the medication prior to baseline visit
* Known intolerance, hypersensitivity or lack of response to duloxetine as judged by the investigator
* A history of treatment resistant depression (defined as 2 or more failed lifetime trials of antidepressant medication as judged by the investigator)
* Currently undergoing psychotherapy that was initiated within the past 3 months
* Significant medical condition that would contraindicate the use of duloxetine or that is untreated and would need urgent attention (as determined by treating physician)
* Medical conditions that would significantly affect absorption, distribution, metabolism, or excretion of duloxetine
* Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
* Any clinically significant deviation from the reference range in clinical laboratory test results as judged by the investigator
* Pregnancy (or female of child-bearing age not using adequate contraception) or lactation
* A positive β-hCG test at enrolment
* Involvement in the planning and conduct of the study
* Previous enrolment or randomisation of treatment in the present study
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
>= 50% improvement in Montgomery-Asberg Depression Rating Scale (MADRS) Scores (MADRS Response) | 12 weeks

SECONDARY OUTCOMES:
MADRS remission | 12 weeks
Credibility and Expectancy Scale (CES) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybook Health Sciences Centre, Toronto, Ontario, Canada